CLINICAL TRIAL: NCT02747134
Title: Combining Emotion Regulation and Mindfulness Skills for Preventing Depression Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/07/178/2678
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Emotion Regulation and Mindfulness skills (Experimental): A 10 week intervention including emotion regulation and mindfulness skills from dialectical behavioral therapy (DBT) was delivered.
  Interventions: Behavioral: Emotion Regulation and Mindfulness skills
- Psychoeducation (Active Comparator): Psychoeducation consisted of 5 session in which basic information about depressive symptoms and how to prevent depression relapse was given.
  Interventions: Behavioral: Emotion Regulation and Mindfulness skills

INTERVENTIONS:
Behavioral: Emotion Regulation and Mindfulness skills

SUMMARY:
In the present study researchers aim to investigate the effectiveness of an intervention combining emotion regulation and mindfulness skills in a single 10-week program. A total of 75 individuals with major depressive disorder (MDD) diagnosis in complete or partial remission participated in this randomized controlled trial (RCT) comparing an intervention including emotion regulation and mindfulness skills (ER+M) with a psychoeducative program. After treatment, participants were followed for a 1-year period. Researchers results indicate that ER+M was not more effective than the treatment used with the control group in preventing depression relapse. Participants allocated to the ER+M group showed a significant decrease on global psychiatric symptoms, whereas those in the control group did not. Further studies are needed in order to better determine the combined effects of mindfulness and behavioral activation.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* having a former MDD diagnosis in complete or partial remission at the time of the study as indicated by the major depressive section of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) and scores below 17 on the Hamilton Depression Rating Scale (HSRD)
* having the last major depressive episode between 18 and 2 months prior to the study
* having at least two previous depressive episodes
* patients could continue pharmacological treatment on condition that it remained stable for at least the last two months before entering the study.

Exclusion Criteria:

* DSM-IV-TR criteria for current MDD or any other affective disorder
* DSM-IV-TR criteria for alcohol or drug dependence, schizophrenia or psychotic disorders
* DSM-IV-TR criteria for personality disorders; severe physical conditions such as organic brain syndrome or neurological disease; mental retardation or cognitive impairments
* having received any psychotherapy including cognitive-behavioral therapy in the past
* changes in the pharmacological treatment during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 1 year

REFERENCES:
- [Derived] Elices M, Soler J, Feliu-Soler A, Carmona C, Tiana T, Pascual JC, Garcia-Palacios A, Alvarez E. Combining emotion regulation and mindfulness skills for preventing depression relapse: a randomized-controlled study. Borderline Personal Disord Emot Dysregul. 2017 Jul 5;4:13. doi: 10.1186/s40479-017-0064-6. eCollection 2017. PMID 28690851